CLINICAL TRIAL: NCT02942095
Title: A Phase I Study of Ixazomib and Erlotinib in Advanced Solid Tumor Patients
Brief Title: Study of Ixazomib and Erlotinib in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0688; NCI-2016-01931 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumors
Keywords: Advanced Solid Tumors; Metastatic cancer; Ixazomib; MLN9708; Erlotinib; Erlotinib hydrochloride; OSI-774; CP358774; Tarceva
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ixazomib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Group - Ixazomib + Erlotinib (Experimental): Dose Escalation Phase: Participants take Ixazomib capsules by mouth on Days 1, 8, and 15 of each 28 day cycle starting with Dose Level 1.
  Participants take Erlotinib tablets by mouth on Days 1 - 28 of each 28 day cycle.
  Interventions: Drug: Ixazomib; Drug: Erlotinib
- Dose Expansion Group - Non Small Cell Lung Cancer (Experimental): Dose Expansion Phase : Participants take Ixazomib capsules by mouth on Days 1, 8, and 15 of each 28 day cycle at the maximum tolerated dose from Dose Escalation Phase.
  Participants take Erlotinib tablets by mouth on Days 1 - 28 of each 28 day cycle.
  Interventions: Drug: Ixazomib; Drug: Erlotinib
- Dose Expansion Group - Pancreatic Ductal Adenocarcinoma (Experimental): Dose Expansion Phase : Participants take Ixazomib capsules by mouth on Days 1, 8, and 15 of each 28 day cycle at the maximum tolerated dose from Dose Escalation Phase.
  Participants take Erlotinib tablets by mouth on Days 1 - 28 of each 28 day cycle.
  Interventions: Drug: Ixazomib; Drug: Erlotinib

INTERVENTIONS:
Drug: Ixazomib — Dose Escalation Phase Starting Dose: Ixazomib 3.0 mg on Days 1, 8, and 15 of a 28-day cycle.
  Dose Expansion Phase: Maximum tolerated dose from Dose Escalation Phase
  Other Names: MLN9708
Drug: Erlotinib — Dose Escalation and Dose Expansion Phase: Erlotinib 150 mg by mouth on Days 1 - 28 of a 29 day cycle.
  Other Names: Erlotinib Hydrochloride; OSI-774; CP358774; Tarceva

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of ixazomib and erlotinib that can be given to patients with advanced solid tumors. The safety of these drugs will also be studied.

This is an investigational study. Erlotinib is FDA approved and commercially available to treat non-small cell lung cancer, but its use in advanced solid cancer is considered investigational. Ixazomib is FDA approved. The study doctor can explain how the study drugs are designed to work.

Up to 36 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of ixazomib and erlotinib based on when you join this study. Up to 4 dose levels of ixazomib will be tested. Up to 18 participants may be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ixazomib is found.

All participants will receive the same dose of erlotinib.

Once the highest tolerable dose is found, up to 18 participants will be enrolled at that dose level as an expansion group.

The dose of the study drug combination that you receive may be lowered if you have intolerable side effects.

Study Drug Administration Each study cycle is 28 days.

You will take ixazomib capsules by mouth on Days 1, 8, and 15 of each cycle.

You will take erlotinib tablets by mouth on Days 1-28 of each cycle.

You should swallow ixazomib capsules whole with 8 ounces (1 cup) of water. Each capsule should be swallowed separately with a sip of water. You should also swallow erlotinib tablets whole with water. You should take the ixazomib and erlotinib doses at the same time.

Do not break, chew, or open the capsules or tablets. Each dose should be taken on an empty stomach, at least 1 hour before or 2 hours after a meal. If you miss a dose, take it as soon as you remember, as long as the next scheduled dose is at least 72 hours (ixazomib) or 12 hours (erlotinib) away. You should not take a double dose to make up for a missed dose. If you vomit after taking a dose, wait until the next scheduled dose. Do not take an additional dose.

Your dose of study drug may be changed and/or you may be given drugs to help control the side effects.

Study Visits:

Cycle 1:

Week 1:

* You will have a physical exam.
* Blood (about 6 teaspoons) will be drawn for routine tests and to check your liver and kidney function.
* If you can become pregnant, leftover blood (about 1 teaspoon) and/or urine will be collected for a pregnancy test.
* During Days 1, 2, 3, 5, and 8, blood (about 1-3 teaspoons) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

Week 2:

°Blood (about 6 teaspoons) will be drawn for routine tests and to check your liver and kidney function.

Week 3:

* You will have a physical exam.
* Blood (about 6 teaspoons) will be drawn for routine tests and to check your liver and kidney function.

Cycle 2 and Beyond:

Week 1:

* You will have a physical exam.
* Blood (about 6 teaspoons) and urine will be collected for routine tests. The blood sample will also be used for liver and kidney function tests.
* If you can become pregnant, part of the routine blood or urine test will be used for a pregnancy test. To continue on this study, you must not be pregnant.

Week 4:

* You will have a physical exam.
* Blood (about 6 teaspoons) will be drawn for routine tests and to check your liver and kidney function.
* On Day 28 of each cycle, if the doctor thinks it is needed, you will have an EKG.
* At the end of every other cycle (Cycles 2, 4, 6, and so on), you will have imaging scans (either CT scans or MRI) performed to check the status of the disease.

If you have side effects or abnormal test results while on study, you may be asked to return to the clinic for more tests until the side effects or abnormal test results improve.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, if you develop new health problems, or if you are no longer able to follow study directions.

Your participation on the study will be over after the end-of-study visit.

End of Study Visit:

Within 30 days after your last dose of the study drugs, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 6 teaspoons) will be drawn for routine tests and to check your liver and kidney function.
* Urine will be collected for routine tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy or that has relapsed after standard therapy or has no standard therapy that increases survival by at least three months.
2. All prior treatment- related toxicities must be CTCAE (Version 4.0) less than or equal to Grade 2 (except alopecia) at the time of screening however clinically relevant AEs that will impact on the ADE of the study drugs or safety of the subject must have resolved to Grade 1 or better.
3. Adequate baseline organ function defined as following: Absolute neutrophil count greater than or equal to 1.5 x 109 cells/L, hemoglobin greater than or equal to 8.0 g/dL, platelets greater than or equal to 75 x 109/L, creatinine less than or equal to 1.5 X upper limit of normal (ULN) with calculated creatinine clearance greater than 30 ml/min, total bilirubin less than or equal to 1.5 X ULN, AST(SGOT) and/or ALT(SGPT) less than or equal to 3 XULN.
4. 18 years of age or older.
5. Life expectancy of at least 3 months in the opinion of investigator.
6. Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
7. Measurable disease as defined by RECIST criteria (Version 1.1).
8. Patients with Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
9. Having archival paraffin tissue is ideal for the correlative study but it is not mandatory.
10. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Female patients who: Are postmenopausal for at least 1 year before the screening visit, OR Are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods]), And latex or non-latex condom with or without a spermicidal agent, Diaphragm with spermicide; Cervical cap with a spermicide; Sponge with a spermicide
12. Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following: a) Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR b) Latex or non-latex condom with or without a spermicidal agent, Diaphragm with spermicide; Cervical cap with a spermicide; Sponge with a spermicide.
13. Inclusion Criteria for dose expansion cohort: Non-small cell lung cancer: 1) We will enroll non-small cell lung cancer patients with documented EGFR mutation who failed treatment with anti-EGFR therapy (e.g. erlotinib or afatinib) and tested negative for EGFR T790M mutation. We will allow patients with positive EGFR T790M mutation if they have progressed on third generation anti-EGFR therapy (e.g. CO-1686 or AZD9291) or medically not suitable/candidate for the third generation anti-EGFR therapy. Failure from anti-EGFR therapy will be defined as progressive disease by RECIST (Version 1.1) after at least two months of therapy. We plan to enroll up to 9 patients in this cohort.
14. Pancreatic ductal adenocarcinoma: 1) Pancreatic ductal adenocarcinoma patient with KRAS point mutation at codon G12 or G13. Since KRAS mutation is present in more than 90% of pancreatic cancer with 98% of the mutation found at codon 12, we expect majority of patients with pancreatic ductal adenocarcinoma will be eligible for the study. We plan to enroll up to 9 patients in this cohort. In addition to the above inclusion criteria, first 5 patients from both non-small cell lung cancer and pancreatic ductal adenocarcinoma patients will need to agree to mandatory pre- and post-treatment tumor biopsies.

Exclusion Criteria:

1. Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
2. Radiotherapy completed within 2 weeks prior to treatment initiation. Radiotherapy completed >2 weeks prior to treatment initiation is allowed if all procedure-related toxicities resolved per inclusion #2.
3. Patient who were receiving prior therapy will require wash out period of either more than 2 weeks or more than 5 half-lives whichever shorter.
4. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
5. Current use of a prohibited medication.
6. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. If these were treated and clinically stable for 4 weeks, patient can be considered for the trial.
7. Patient who is on strong inducer/inhibitor of CYP3A needs to be off the medication prior to treatment initiation unless it is medically necessary for the patient.
8. Female patients who are lactating or have a positive serum pregnancy test suggestive of pregnancy and not as a tumor marker during the screening period. If pregnancy is tested positive, treating physician will further investigate if the patient is pregnant or not. Treating physician may consider repeating the serum beta-hCG at next follow up visit or refer patient to OB/GYN for further evaluation.
9. Major surgery within 14 days before enrollment.
10. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
11. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
12. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
13. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
14. Patient has greater than or equal than Grade 2 peripheral neuropathy, or Grade 1 with pain on clinical examination during the screening period.
15. Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ixazomib and Erlotinib in Advanced Cancer Participants | 28 days
  MTD defined by dose limiting toxicities (DLTs) that occur during the first cycle.
  Dose limiting toxicity (DLT) defined as
  1. Any Grade 3 or 4 non-hematologic toxicity as defined in the NCI CTCAE.
  2. Any Grade 4 hematologic toxicity lasting two weeks or longer (as defined by the NCI-CTCAE), despite supportive care.
  3. Grade 4 nausea, vomiting or diarrhea > 5 days despite maximum anti-nausea regimens.

SECONDARY OUTCOMES:
Tumor Response of Ixazomib and Erlotinib in Participants with Non Small Cell Lung Cancer | 8 weeks
  Tumor response of this combination per RECIST version 1.1.
Tumor Response of Ixazomib and Erlotinib in Participants with Pancreatic Ductal Adenocarcinoma | 8 weeks
  Tumor response of this combination per RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org